

#### **BULLYDOWN**

# ASSENT FORM FOR CHILDREN AGES 11 - 14

PROJECT TITLE: BullyDown

FUNDER: National Institute of Child Health and Human Development

PRINCIPAL INVESTIGATOR NAME: Dr. Michele Ybarra Telephone: (877) 302-6858, extension 801

Email: Michele@InnovativePublicHealth.org

Additional Contact: Dr. Dorothy Espelage

Telephone: 217-766-6413 Email: espelage@unc.edu

- We are asking you to take part in a test of BullyDown, a program to help kids stop bullying.
- You will get 3-5 text messages every day for about 8 weeks. Text messages will be about how to stop bullying.
- We will ask you to do 3 surveys: One at the beginning, one at the end of the program, and one 3 months later. To be in the program, you need to complete the first suvey.f
- If you take part, we might send you a message or ask you a question that makes you feel uncomfortable.
- There may be no benefit to you to take part, but your feedback about being in the program will help us build a better program for youth about bullying in the future.

## **Background**

BullyDown is a bullying prevention program that is delivered by text messaging. We will send about 3-5 messages to your cell phone each day for about 8 weeks. The messages will talk about things like communication, things kids think about bullying, the way bullying can make kids feel, and some ideas about how to deal with bullying if it happens.

This research study is sponsored by the National Institutes of Health.

## **Procedures**

You are one of about 200 middle school students who we are getting assent from to take part in a test of BullyDown.

We are testing two different text messaging programs to stop bullying. We do not know which one works better. You will be put in one group or the other randomly. This means you will be assigned to one program or the other by chance alone, like rolling dice. We will not tell you or your guardians/parents which program you are assigned to until after everyone has finished the program.

If you take part in the research study, here is what we are asking you to do:



Expires: 04/04/2024

Complete three online surveys: One at the beginning of the study, one at the end of the study, and one three months after the study.

- Read messages every day for about 8 weeks.
- Every week, we will send a couple of text messages with questions about your experiences in the program and ask you to answer via text messaging.
- We may ask you if you want to do a phone interview with research staff about your experience in the program at the end of the study.

You also might be matched with a "Text Buddy." This person is another middle school student in this study that you will be able to text message about the things that you are learning in the program. You also may have access to "Forever Friend," which is a feature that will send you a happy message whenever you text it.

### **Incentives**

You will get \$15 for each of the three surveys that you do. If you do all three surveys, you will get \$45 after completing the third survey (three months after the intervention ends). It will be sent as an Amazon gift card.

### **Risks and Discomforts**

You can choose to be in the study or not. If you decide not to be in the study, that is OK. You can choose to stop being in the study at any time, even if you have already started.

It is possible that we will send you a message or ask you a question that makes you feel weird or you do not like. If so, you can skip it. If someone sees your cell phone screen, they may see messages from the program and know you are learning about bullying. It also is possible that your privacy will be broken if you or your Text Buddy share the messages you send to each other. We will ask both of you not to but we cannot promise this will happen. Your buddy will be from a different school.

### **Benefits**

We do not know if being in the study will help you. But, your feedback will help us design a better program about bullying for middle school students in the future.

# Rights of Refusal and Withdrawal

It is your choice to take part in the study or not. If you decide not to be in the study, nothing bad will happen. Also, you may change your mind and stop taking part at any time.

If, at any time, you no longer want to be in the study, please contact us to let us know by emailing us at Michele@InnovativePublicHealth.org or texting us at: (714) 252-4660.

Your time in the study may also stop at any time for any reason, such as, the sponsor or the study investigator decides to stop the study.

#### **Confidentiality**

We will not tell your parents your answers in the study.

We will keep a copy of your answers after the study ends so that we can look at them later. We will only share research data where we have removed anything that we think would show your

Pearl RB
Protocol: 21-CIPH-IPI-GPHty There still

Protocol: 21-CIPH-Indepartity. There still may be a small chance that someone could figure out that the information is Expires: 04/05/2023 Expires: 04/04/2024about you. Such sharing includes:

- Publishing results in a book or journal.
- Adding results to a Federal government database.
- Using research data in future studies, done by us or by other scientists.
- Representatives at the Department of Health and Human Services and Pearl IRB also may request access to the study data.

To help us protect your privacy, we have obtained a Certificate of Confidentiality from the National Institutes of Health. This Certificate means that we can keep your information private even if we get a court order telling us to share your information. We will use this Certificate to fight demands for your information unless you tell us you want us to share the information. But in the unlikely event that you tell us that you are being harmed or harming others, then under applicable law we may be required to report this information to the appropriate authorities.

### **Questions and Contact Numbers**

If you have questions about the study, or any concerns about the study questions, please contact:

- Dr. Michele Ybarra toll-free at 1-877-302-6858 ext. 801 or Michele@InnovativePublicHealth.org
- Dr. Dorothy Espelage, via email at espelage@unc.edu or phone at 217-766-6413.

If you have questions about your rights as a participant in this study, or if you feel that you have been harmed in any way by taking part in this study, please contact Pearl IRB:

• By mail: Study Subject Adviser Pearl IRB 29 East McCarty Street, Suite 100 Indianapolis, IN 46225 or call: 317-899-9341 or by email: info@pearlirb.com

By clicking yes below, it means that **you agree** to take part in this research study. If you click no below, it means that you **do <u>not</u> agree** to take part in this research study. Yes

No